CLINICAL TRIAL: NCT01411423
Title: Special Drug Use Investigation of Nexavar (Unresectable or Advanced Renal Cell Carcinoma)
Brief Title: Nexavar Post-marketing Surveillance for Renal Cell Carcinoma in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15038; NEXAVAR-RCC-02 (Other: Company Internal)
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Carcinoma, Renal Cell
Keywords: Nexavar; Unresectable or advanced renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Patients who have received Nexavar for unresectable or advanced RCC.

SUMMARY:
This study is a regulatory post-marketing surveillance in Japan, and it is a local prospective and observational study of patients who have been administered with Nexavar for unresectable or advanced renal cell carcinoma (RCC). The objective of this study is to assess safety and effectiveness of Nexavar under real-life practice conditions. This study is an all case investigation of which the enrollment period is 15 months, and all patients who received Nexavar will be recruited and followed one year since starting Nexavar administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received Nexavar for unresectable or advanced renal cell carcinoma

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is all cases investigation of which the enrollment period is 15 months, and all patients who received Nexavar for unresectable or advanced RCC will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 3305 (Actual)
Dates: Start 2008-04-18 (Actual); Primary Completion 2012-03-16 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions and serious adverse events in subjects who received Nexavar | After Nexavar administration, up to 1 year

SECONDARY OUTCOMES:
Incidence of adverse drug reactions in subpopulation in a variety of baseline data [such as demographic data, concomitant disease, medical history data, clinical staging, etiology of HCC, Eastern Cooperative Oncology Group-Performance Status (ECOG-PS)] | After Nexavar administration, up to 1 year
Effectiveness evaluation assessment [overall survival, response rate, stable disease rate, progression disease rate] by investigator-determined overall best response [according to the General rule for clinical and pathological studies on RCC] | After Nexavar administration, up to 1 year
The status of therapy with Nexavar [duration of treatment, daily dose] | After Nexavar administration, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Derived] Inamoto T, Azuma H, Tatsugami K, Oya M, Adachi M, Okayama Y, Sunaya T, Akaza H. Real-world use of sorafenib for advanced renal cell carcinoma patients with cardiovascular disease: nationwide survey in Japan. Expert Rev Anticancer Ther. 2020 Jul;20(7):615-623. doi: 10.1080/14737140.2020.1773805. Epub 2020 Jun 16. PMID 32441582